CLINICAL TRIAL: NCT06525415
Title: Foot Perfusion by Dynamic Contrast Enhanced MRI in Patients With Peripheral Artery Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Other Study IDs: 2024ZW001
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Peripheral Arterial Disease; Perfusion
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Dynamic Contrast Enhanced Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PAD group: patients of peripheral artery disease who underwent endovascular treatment
  Interventions: Diagnostic Test: DCE MRI

INTERVENTIONS:
Diagnostic Test: DCE MRI — the recruited patients should complete pre- and post-operative DCE MRI workshops

SUMMARY:
We investigate the peri-operative foot perfusion through dynamic contrast enhanced MRI in patients with peripheral artery disease

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old;
* PAD patients with Fontaine grade II-IV or Rutherford grade 2-6 and underwent a successful revascularization;
* Patients completed both pre- and post-operative MRI workups;
* Patients signed the informed consent form and be able to complete the clinical follow-up for 1 months.

Exclusion Criteria:

* Patients has participated in other clinical studies;
* Patients with Heart failure (NYHA III/IV)/right to left shunt heart disease/ severe aortic and mitral insufficiency/acute coronary syndrome/malignant arrhythmia/severe pulmonary hypertension (pulmonary artery pressure at least 90 mmHg)/moderate to severe renal insufficiency (creatinine clearance rate<60 ml/min)
* Any allergic constitution;
* Pregnancy and childbirth;
* Life expectancy<12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with peripheral artery disease, who had a successful endovascular treatment and completed both pre- and post-operative MRI workups
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
preoperative perfusion parameters | Between Aug.1 2024 and OCT.31 2024
  preoperative perfusion parameters by dynamic contrast-enhanced (DCE) magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
ankle brachial index | Between Aug.1 2024 and OCT.31 2024
clinical success | Between Aug.1 2024 and NOV.30 2024
survival | Between Aug.1 2024 and NOV.30 2024

IPD SHARING:
Plan to Share IPD: Undecided